CLINICAL TRIAL: NCT02659306
Title: The Effect of Metformin on HIV Reservoir Size in Non-diabetic Antiretroviral Therapy (ART) Treated Participants: the Lilac Study
Brief Title: Metformin Immunotherapy in HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Jean-Pierre Routy, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTNPT027
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): Assessment will be done at the baseline, during and after 12 week of metformin use.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin hydrochloride is a white to off-white crystalline compound formulated as tablets for oral consumption; tablets contain 500 mg, 850 mg, or 1000 mg of metformin hydrochloride. Only 500 mg and 850 mg tablets will be used for this study.
  Other Names: Glucophage

SUMMARY:
Anti-HIV drugs cut down the number of serious infections that people with HIV get. However, some subjects taking anti-HIV drugs do not achieve adequate cluster of differentiation 4 (CD4) recovery and decrease in elevated cluster of differentiation 8 (CD8) cells. Such patients with a low CD4/CD8 ratio remain at risk for developing acquired immune deficiency syndrome (AIDS) and non-AIDS-related complications. Two of the most important factors associated with low CD4/CD8 ratio include: the persistence of HIV on ART and inflammation.

Metformin, the most widely used medication to treat type 2 diabetes, is well tolerated with minimal side effects. It has been linked to anti-aging and weight reducing properties in non-diabetic persons. Because of its ability to improve immune functions, metformin could be a promising addition to ART in HIV patients. It is also reported to change the composition of microbes in the gut which may improve inflammation.

PURPOSES OF THE STUDY

The purposes of this study are to find out if:

1. metformin can be combined with anti-HIV drugs to reduce the amount of hidden virus in the body;
2. metformin can be combined with anti-HIV drugs to improve immune function.
3. metformin can be combined with anti-HIV drugs to impact CD4 T cell count and CD4/CD8 T cell ratio during treatment and after its discontinuation
4. metformin can change the composition of the bacteria in the gut which may improve inflammation.

For this purpose, the investigators will add metformin at the usual antidiabetic dose for 12 weeks for patients receiving stable ART, having a CD4/CD8 ratio below 0.7.

Approximately 22 participants will be enrolled in this study at the Chronic Viral Illness Service of the McGill University Health Centre, the Ottawa Hospital and the Maple Leaf Medical Clinic (Toronto). This study will last about 24 weeks; metformin treatment will be for 12 weeks. In order to be eligible for the study, the participants must be 18 years of age or older, have an undetectable viral load (the quantity of the HIV virus in the blood must be less than 50 copies/ml) for at least 3 months and have a CD4/CD8 ratio of less than 0.7. All participants will also be asked to give blood and stool samples and optional colon mucosal biopsy samples (before and after metformin supplementation) to study the size of the viral reservoir and the amount of T cell activation and changes in gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected male or female adults greater than or equal to 18 years of age
2. HIV-1 infected adults successfully treated with ART for at least 3 years (the time necessary to establish a stable reservoir)
3. Individuals on a stable ART regimen for at least 3 months, with plasma viral load below the level of detection and with a CD4/CD8 ratio ≤ 0.7
4. Non-diabetic (HbA1c < 5.9%) and pre-diabetic individuals (HbA1c between 6.0 and ≥ 6.4%), as defined by their glycosylated hemoglobin levels
5. Able to understand and sign the informed consent form prior to screening

Exclusion Criteria:

1. Individuals with a known hypersensitivity/allergy to the metformin
2. Individuals who are actively participating in an experimental therapy study or who have received experimental therapy within the last 6 months
3. Individuals who are suffering from severe systemic diseases (uncontrolled hypertension, chronic renal failure), or active uncontrolled infections
4. Individuals having diabetes mellitus (HbA1c ≥ 6.5 %) as defined by the Canadian Clinical Practice Guidelines for the Prevention and Management of Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09; Primary Completion 2018-08-14 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Decrease in the size of the HIV reservoir | 12 weeks

SECONDARY OUTCOMES:
Change in the percentage of activated CD8 T-cells | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Routy, MD; FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Chronic Viral Illness Service, McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Background] Routy JP, Mehraj V, Cao W. HIV immunotherapy comes of age: implications for prevention, treatment and cure. Expert Rev Clin Immunol. 2016;12(2):91-4. doi: 10.1586/1744666X.2016.1112269. Epub 2015 Dec 2. PMID 26629806
- [Background] Lu W, Mehraj V, Vyboh K, Cao W, Li T, Routy JP. CD4:CD8 ratio as a frontier marker for clinical outcome, immune dysfunction and viral reservoir size in virologically suppressed HIV-positive patients. J Int AIDS Soc. 2015 Jun 29;18(1):20052. doi: 10.7448/IAS.18.1.20052. eCollection 2015. PMID 26130226
- [Background] Vyboh K, Jenabian MA, Mehraj V, Routy JP. HIV and the gut microbiota, partners in crime: breaking the vicious cycle to unearth new therapeutic targets. J Immunol Res. 2015;2015:614127. doi: 10.1155/2015/614127. Epub 2015 Feb 22. PMID 25759844
- [Background] Dagenais-Lussier X, Mouna A, Routy JP, Tremblay C, Sekaly RP, El-Far M, Grevenynghe Jv. Current topics in HIV-1 pathogenesis: The emergence of deregulated immuno-metabolism in HIV-infected subjects. Cytokine Growth Factor Rev. 2015 Dec;26(6):603-13. doi: 10.1016/j.cytogfr.2015.09.001. Epub 2015 Sep 8. PMID 26409789
- [Derived] Routy JP, Isnard S, Mehraj V, Ostrowski M, Chomont N, Ancuta P, Ponte R, Planas D, Dupuy FP, Angel JB; Lilac Study Group. Effect of metformin on the size of the HIV reservoir in non-diabetic ART-treated individuals: single-arm non-randomised Lilac pilot study protocol. BMJ Open. 2019 Apr 20;9(4):e028444. doi: 10.1136/bmjopen-2018-028444. PMID 31005944
- See also: The Canadian HIV Trials Network — http://www.hivnet.ubc.ca/home/